CLINICAL TRIAL: NCT06573086
Title: Towards Personalized Exercise: Identifying the Determinants of Individual Variation in Repeated Resistance Training (TraDeRe) and Examining Transferability of Responsiveness Between Resistance Training and Endurance Training
Brief Title: Resistance Training, Detraining, and Retraining Study 2024 (TraDeRe2024)
Acronym: TraDeRe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Juha Ahtiainen, Associate Professor, University of Jyvaskyla
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1394/13.00.04.00/2023
Record Dates: First submitted 2024-07-29; First posted 2024-08-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophy; Exercise Training; Skeletal Muscle Atrophy; Healthy
MeSH Terms: conditions — Hypertrophy; Muscular Atrophy | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High responders (n=30) (Experimental): This group consists of participants with the highest increase in skeletal muscle hypertrophy of m. vastus lateralis in response to the initial 12 weeks of RT (Intervention I).
  Interventions: Other: Resistance Training
- Moderate responders (n=30) (Experimental): This group consists of participants with the moderate increase in skeletal muscle hypertrophy of m. vastus lateralis in response to the initial 12 weeks of RT (Intervention I).
  Interventions: Other: Resistance Training
- Low Responders (n=30) (Experimental): This group consists of participants with the lowest increase in skeletal muscle hypertrophy of m. vastus lateralis in response to the initial 12 weeks of RT (Intervention I).
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — 12-week resistance training
  Other Names: Exercise Training

SUMMARY:
The goals of our research project are to identify factors explaining inter-individual variation in responses to resistance training (RT) and the baseline determinants underlying an individual's sensitivity to respond to RT. Moreover, investigators aim to assess whether a responsiveness to RT predicts responsiveness to endurance training (ET). Thus, investigators aim to gain a deeper understanding of exercise adaptation processes. The main questions investigators aim to answer are:

* Can the physiological responses of one RT intervention be extrapolated to a subsequent RT intervention?
* If so, what are the mechanisms underlying differing skeletal muscle growth responses in low, and high responders of skeletal muscle hypertrophy?
* If so, do the low responders of skeletal muscle growth respond more favourably when the amount of RT is increased?
* Are the high, moderate, and low responders of RT also the highest, moderate, and lowest responders to ET?

To examine these main research questions, high (n=30), low (n=30), and moderate (n=30) responders of skeletal muscle growth in response to RT (intervention I, NCT05874986) are reallocated into a subsequent 12-week RT intervention (intervention II) after a detraining period. A subgroup of these participants (n=10) will engage in a 6-week control period before starting the second RT period. Additionally, after intervention II, participants will participate in an ET intervention, lasting 6 weeks.

In this intervention II, reallocated participants will be:

* Resistance training with supervision for 12 weeks
* Consuming deuterium oxide for the assessment of muscle protein synthesis
* Consuming D3-3-methylhistidine for the assessment of acute muscle protein breakdown
* Consuming D3-creatine for the examination of whole-body skeletal muscle mass
* Providing a spot urine sample six (6) times, and urine collection for 24 hours performed twice
* Providing saliva samples (30-32 in total) for the assessment of body water enrichment of deuterium
* Providing a muscle biopsy four or five (4-5) times during the study
* Providing a blood sample fourteen (14) times during the study
* Assessed for body composition and body volume four or five times (4-5) during the study
* Participating in muscle size, maximal dynamic strength and TMS measurements four or five (4-5) times during the study
* Asked to answer questionnaires related to e.g. stress, physical activity, sleep, perceived exertion, and diet
* Participating in recovery measurements before and after the second-to-last and the last RT bout, and once in the days between these RT bouts, consisting of six (6) body volume measurements and six (6) maximal voluntary isometric contraction (kg) tests using horizontal leg press for the assessment of neuromuscular recovery
* Participating in an acute resistance exercise (RE) after the 12-week RT intervention.

Furthermore, in the ET intervention, participants will be:

* Participating in a familiarization session and resting electrocardiograph measurements before the intervention
* Participating in endurance testing consisting of body composition, movement economy, and incremental RAMP testing before and after ET intervention
* Endurance training with supervision for 6 weeks, three times a week.

DETAILED DESCRIPTION:
While the diverse health and performance benefits of resistance training (RT) are widely recognized, some individuals demonstrate notably divergent responses to RT intervention. This phenomenon is termed inter-individual response variation to RT. However, despite the prevalence of these research findings, the precise underlying mechanisms contributing to these differential RT responses remain ambiguous. Finally, it is currently unknown whether a responsiveness to RT predicts responsiveness to ET within the same set of participants, as this area of research is critically understudied.

Investigators aim to investigate the cellular, molecular, and neuromuscular mechanisms behind the plausible RT response variability intra- and inter-individually, using trial-to-trial, i.e. resistance training, detraining, and retraining design. Moreover, as the impact of diverse polygenic effects on RT responsiveness is yet to be determined, investigators will employ a multi-OMIC (genomic, epigenomic, transcriptomic, proteomic, and metabolomic) approach to unravel previously unknown denominators of RT responsiveness. Finally, numerous environmental factors, e.g. nutrition, stress, sleep, and physical activity are monitored during the study to assess the effects of non-physiological mechanisms on RT response variability.

In our study, 362 healthy male and female participants in total started in the study and were destined to undergo an RT period of 12 weeks in two separate periods (intervention I refers to NCT05874986). Then, a subset of the participants from intervention I will be reallocated into intervention II based on the magnitude increase of m. vastus lateralis (VL) cross-sectional area (CSA) assessed by ultrasound using extended-field-of-view mode. Similar to intervention I, intervention II will be performed in separate periods similarly to the data collection I and II of intervention I to first accumulate approximately 32 weeks of detraining for both cohorts, after which 12 weeks of RT is performed.

Moreover, a subset (n=30) of the participants aged 40-50 from intervention I not selected for intervention II have a chance to take part in a 10-week home training sub-study. These participants will be randomized to a non-training control group (n=15) and a home training group (n=15). The home training group will carry out a 10-week RT period utilizing muscle-strengthening activities in their home. This sub-study investigates how minimally supervised RT executed at home after supervised gym RT can maintain muscle strength and size compared to non-training. Home training is flexible, time-saving, and inexpensive. It is also done twice weekly using safe and effective training protocols and movements. Home-based training includes pistol squat, reverse nordic, push up, and bent-over row, and bicep curl exercises. To achieve progression, the total load will be increased by increasing the number of repetitions per set, and/or increasing the load by using a progression from easier to more difficult techniques and/or by adding resistance bands, which will be provided to participant's free of charge for the duration of the study. Participants will be contacted regularly to ensure motivation and adherence to home exercise. All the participants in this sub-study, as well as the other participants not selected for intervention II are offered a self-directed, non-supervised 7-week RT period with a similar design as in intervention I with access to our gym located in our Faculty's building. VL CSA, horizontal leg press 1 repetition maximum, and body composition will be assessed before and after home training and self-directed RT for each participant.

In intervention II, participants will be performing RT similarly to intervention I. However, for the last 5 weeks of the intervention, RT volume will be increased by 40 % for the lower body exercises to assess the impact of RT volume increment on RT responses. After 12 weeks of RT, an experimental RT session will be conducted to assess the acute physiological responses to resistance exercise. The experimental session will consist of five heavy sets of both horizontal leg press and leg extension exercises. During the last RT week, participants will engage in recovery measurements before and after the second-to-last and the last RT bout, and once during the days between these two bouts. After 12 weeks of RT, participants will be performing an additional acute resistance exercise session. All the participants NOT selected for intervention II are able to participate in a self-directed, 6-week RT period with measurements before and after this period. These measurements include body composition, muscle size (VL CSA and muscle thickness of elbow flexors) and muscle strength (dynamic 1RM of horizontal leg press and barbell scott curl) assessments. A subgroup of the participants (n=10) will engage in a control period of 6 weeks in duration, before the onset of RT.

After the intervention II, participants will begin a washout period lasting approximately 16 weeks (± 2), during which participants are advised to abstain from RT and ET. After a washout period, participants will participate in the familiarization measurements regarding the ET intervention. In familiarization, participants are measured with an electrocardiogram (ECG), after which a medical doctor will evaluate the resting ECG results to verify the eligibility of each participant. Moreover, participants will be habituated to movement economy testing by performing 3x3 min low-intervals with loads of 30-55-80 watts for females and 50-80-110 watts for males, respectively, and other included measurements. After familiarization and eligibility assessment, baseline measurements will be conducted the following week. Baseline measurements include body composition and volume assessment with a 3D optical body scanner, a 4 x 4 minute movement economy test with individualized, progressive loads determined in the familiarization (last load near the aerobic threshold). Movement economy intervals are performed with no rest in between. Finally, a maximal oxygen uptake (VO2max) will be measured breath-by-breath with an incremental RAMP test. The starting intensity will be 30 watts for both males and females, and the intensity will be increased by 30 and 25 watts per minute for males and females, respectively. The RAMP test will be performed with a self-selected cadence above 60 rounds per minute (rpm). When participants fail to maintain a cadence over 60 rpm second time, after one warning and despite heavy encouragement, the RAMP test will be terminated. All the testing will be performed using a bicycle ergometer. Heart rate, heart rate variability (HRV), expired gas analysis, arterial oxygen saturation, power output, stroke volume and cardiac output will be monitored continuously during the tests. Perceived exertion is assessed with a modified RPE scale of 0-10 after each movement economy interval and RAMP test. Blood lactate, blood glucose and hemoglobin concentrations are also measured after each movement economy interval and at the end of the RAMP test.

Endurance exercise is programmed based on the guidelines by the American College of Sports Medicine. During weeks 1-2, 45 minutes of low-intensity (= near the first ventilatory threshold) steady-state cycling is performed. In weeks 3-4, 50 minutes of cycling is performed, during which every other session includes low intensity cycling and every other session 3 x 10-minute intervals (with 4-minute rest after each interval) at moderate intensity (= between the first and the second ventilatory thresholds). Finally, in weeks 5-6, 55 minutes of cycling is performed, consisting of 4 x 10-minute intervals (with 3-minute rest after each interval) at a moderate intensity. Participants will be doing endurance exercises in groups of 2-4, and training three times a week at the standardized time of day. At the beginning of ET, appropriate training intensities are verified with blood lactate and the modified RPE scale. Training intensities at the start are decided by two blinded researchers based on the ventilatory thresholds obtained during the RAMP test. Individual training data, including heart rate, HRV, RPE, and wattage, is collected. The wattage is continuously displayed on the screen of the cycle ergometers during sessions to maintain appropriate training intensities. Wattage is increased within and between training sessions according to heart rate, lactate concentration, and modified RPE scale to establish progression. Before the onset of each interval session, a brief low-intensity steady-state warm-up of 7-8 minutes is performed.

In this study, investigators aim to identify several previously unknown molecular determinants that underlie the observed heterogeneity in RT responses. This could significantly increase the understanding of exercise physiology, which can be applied, e.g., in sports medicine, rehabilitation, and sports coaching. Moreover, this study can promote the development of personalized exercise prescriptions as part of health care. Indeed, it is vital to examine whether the same individuals respond similarly or differently to RT and ET at least in the short term. These findings can then be used to adjust individualized training programming not only as a part of health care but also regarding physical performance optimization. Finally, the findings of the study can operate as a foundational work for future research on the topic of RT response heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* healthy (e.g., no diagnosed type 2 diabetes, cardiovascular disease, musculoskeletal disorders, etc.)
* prior participation in intervention I (NCT05874986)

Exclusion Criteria:

* medication affecting the cardiovascular system or metabolism
* metabolic, musculoskeletal, cardiovascular, or other diseases or disorders which may preclude the ability to perform exercise training and testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in m. vastus lateralis (VL) cross-sectional area (CSA) with ultrasound (US) | Baseline (test and retest), week 7, week 13
  VL CSA (cm^2) is determined at mid-thigh using a B-mode axial plane US (Venue Fit R4, GE Medical Systems, USA) with a L4-20t-RS linear-array probe (48,43 mm width) in extended-ﬁeld-of-view mode (6/12 MHz, 39 frames per second).
  Additionally, VL CSA (cm^2) will also be determined at baseline with different US, at mid-thigh using a B-mode axial plane US (model SSD-α10, Aloka, Tokyo, Japan) with a 13 MHz linear-array probe (60 mm width) in extended-ﬁeld-of-view mode (23 Hz sampling frequency). Aloka-US was used in the intervention I, but GE-US in intervention II due to the progressive malfunctioning of Aloka. Therefore, both machines are used in baseline measurements to calculate the plausible inter-US variability.
  The CSA will be measured using the polygon function in ImageJ software. Per each measurement, three images will be analysed from which the average from the two closest ones will be calculated.

SECONDARY OUTCOMES:
Muscle protein synthesis (MPS) with the Combined Oral Stable Isotope Assessment of Muscle (COSIAM) | From baseline to week 7 (6 weeks of RT in duration)
  A baseline saliva sample is collected to determine the deuterium labelling of plasma proteins. Then, participants ingest 3ml/kg deuterium oxide (D2O, 70-Atom%) divided into three boluses and 1 ml/kg top-up dose twice a week throughout the MPS examination period. When muscle proteins are built, the accumulation of deuterium-labelled alanine amino acid in the VL can be used to measure local fractional sarcoplasmic, myofibrillar, mitochondrial, and collagen MPS rates via gas chromatography-pyrolysis-isotope ratio mass spectrometry (GC-Pyrolysis-IRMS). The outcome will be expressed as %/day. 30 mg of VL muscle biopsy is used for MPS analysis. To estimate alanine precursor enrichment (APE), saliva samples are collected before and after each D2O drink consumption and 24 and 48 hours after the 3 x bolus to monitor body water enrichment via thermal conversion elemental analyser (TC/EA)-IRMS. Mass spectrometry analyses will be performed at the University of Nottingham, United Kingdom.
Muscle protein breakdown (MPB) with the Combined Oral Stable Isotope Assessment of Muscle (COSIAM) | Baseline, Week 7
  Before each measurement day, participants ingest 10 mg of stable isotopically labelled D-3-methylhistidine (D-3-MH) dissolved in 50 millilitres of water. When muscle proteins containing D-3-MH are degraded, D-3-MH is released into circulation. As D-3-MH cannot be reused for protein synthesis, D-3-MH can be used as a biomarker for muscle protein breakdown (MPB). The enrichment of labelled D-3-MH is then measured from the blood samples to assess MPB. The outcome will be expressed as the tracer dilution (k) rate of D3-3-MH and measured with repeated plasma sampling. 20-24 hours after the ingestion of D3-3MH, five plasma samples will be collected within three hours, each separated by 45 minutes. Plasma samples will be analysed at the University of Nottingham, United Kingdom.
Change in whole-body skeletal muscle mass (SMM) with the Combined Oral Stable Isotope Assessment of Muscle (COSIAM) | Baseline, Week 7
  First, a baseline urine sample is collected to measure D3-creatinine enrichment. Then, after the bladder is empty, participants consume 30 mg of labelled D3-creatine dissolved in 50 millilitres of water. The amount of D-3 creatine that spills over in urine samples after 24 hours of ingestion will then be used to determine the amount of D-3 creatine retained in the body by 24-hour urine collection. Then, as the amount of creatine-to-creatinine conversion remains similar in the total muscle pool, the comparison of both non-labelled and labelled creatinine can be used to estimate the whole-body muscle creatine pool from the urine samples gathered 48 to 72 hours post-ingestion. This enables the calculation of whole-body skeletal muscle mass with a simple equation and the following outcome will be expressed as kilograms (kg). Urine samples will be analysed at the University of Nottingham, United Kingdom.
Change in muscle thickness (MT) of the elbow flexors after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  MT of m. biceps brachii and m. brachialis is measured using a B-mode axial plane ultrasound (Venue Fit R4, GE Medical Systems, USA) with a L4-20t-RS linear-array probe (48,43 mm width).
Change in lower and upper limb maximal strength after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13,
  Maximal voluntary concentric muscle strength of leg extensors is determined in a horizontal leg press device (David 210) via a one-repetition maximum (1RM) test. Moreover, the maximal voluntary concentric muscle strength of elbow flexors is also measured using barbell bicep curl performed in Scott bench. Maximum strength tests are performed according to the National Strength and Conditioning Association (NCSA) guidelines.
  Both concentric muscle strengths are expressed as kilograms (kg).
Change in corticoreticular excitability after resistance training with transcranial magnetic stimulation (TMS) | Baseline (test and retest), week 7, week 13
  Electrical stimulation of the brachial plexus is performed during rest to elicit the maximum M-wave (M-max) of the biceps brachii. M-max is obtained by increasing the stimulator output intensity until the electromyography (EMG) response plateau. M-max is recorded using surface EMG. Next, single TMS pulses are delivered during tempo-controlled dynamic barbell bicep curls performed with a 30% load of one repetition maximum (1 RM). The TMS pulses are administered when the elbow joint flexion angle reaches 110 degrees. The stimulation intensity will be 100% of the maximum output. The protocol consists of two phases: the first involves four sets of five repetitions, followed by one set of 40 repetitions. Using TMS, investigators analyze the motor-evoked potential (MEP) amplitude, contralateral (cMEPs) and ipsilateral (iMEPs), the iMEP/cMEP amplitude ratio (ICAR), latency, and the silent period, all extracted from the EMG signal.
Change in ribosome biogenesis | Baseline, week 7, week 13
  A portion of the VL muscle biopsies will be used for ribosomal analyses. Ribosome biogenesis and changes in messenger RNA and protein expression will be determined from the muscle biopsy samples by measuring ribosomal RNA and its regulators using real-time quantitative polymerase chain reaction (PCR) and proteomics.
Change in muscle fiber capillarization | Baseline, week 7, week 13
  A portion of the VL muscle biopsies will be used for immunohistochemical analysis. CD56 is used as an antibody for capillaries with a specific secondary fluorophore-labelled antibody. The structural quantification will be performed automatically using an artificial intelligence (AI)SDS PA-based software in Fiji.
Change in muscle fiber cross-sectional area (CSA) during the intervention period | Baseline, week 7, week 13
  A portion of the VL muscle biopsies will be used for immunohistochemical analysis. MANDYS8 antibody is used for staining muscle fiber borders with a specific secondary fluorophore-labelled antibody. Muscle fiber CSA will be quantified using an AI-based software in Fiji.
Change in myonuclear content of the muscle fibers | Baseline, week 13
  A portion of the VL muscle biopsies will be used for immunohistochemical analysis. PCM1 is used as an antibody for myonuclei with a specific secondary fluorophore-labelled antibody. Myonuclear content will be quantified using AI-based software in Fiji.
Change in satellite cell content during the intervention of the muscle fibers | Baseline, week 13
  A portion of the VL muscle biopsies will be used for immunohistochemical analysis. Pax7 is used as an antibody for satellite cells with a specific secondary fluorophore-labelled antibody. Satellite cell content will be quantified using AI-based software in Fiji.
Change in macrophage content of the muscle fibers | Baseline, week 7, week 13
  A portion of the VL muscle biopsies will be used for immunohistochemical analysis of macrophage content with the methods and primary (CD11b, CD206) and fluorophore-labelled secondary antibodies commonly utilized in our laboratory. Macrophage content will be quantified using AI-based software in Fiji.
Changes in anaerobic enzymes | Baseline, week 7, week 13
  Will be measured by Western blotting and Sodium Dodecyl Sulfate Polyacrylamide Gel Electrophoresis (SDS-PAGE).
Changes in sarcoplasmic protein contents | Baseline, week 7, week 13
  Will be measured by Western blotting and SDS-PAGE.
Changes in multiomics during the intervention | Baseline, week 13
  Blood and muscle samples are used for the OMIC analyses. DNA extraction will be performed from blood and muscle samples in our Faculty.
  For genomic analysis, DNA samples will be sent to the Institute for Molecular Medicine Finland to produce single nucleotide polymorphisms using the advanced genotyping array (Illumina Infinium Global Screening Array-24v2.0 BeadChip). Then, quantitative genome-wide polygenic risk score (PRS) will be quantified using known genomic loci. Epigenetic analysis for DNA methylation will be assessed by Illumina's Infinium Methylation EPIC BeadChip (Illumina, San Diego, CA, USA). Transcriptomic profiling will be performed by RNA sequencing. Proteome profiling will be performed using large format difference in-gel electrophoresis (DiGE). Lastly, a high-throughput serum Nuclear Magnetic Resonance (NMR) metabolomics platform will be used for the absolute quantification of serum lipids and metabolite profiles.
Satellite cell isolation | Week 13
  From muscle biopsy samples, satellite cells will be isolated, and fibroblast-free primary satellite cell cultures will be established using the methods recently applied in our laboratory. Cultures of differentiated myotubes can be later utilized in mechanistic studies to examine specific molecular networks revealed by OMIC analyses.
Change in whole body fat mass | Baseline (test and retest), week 7, week 13
  Fat body mass (kg) is measured at morning after overnight fasting by bioimpedance device (InBody 770, Biospace Co. Seoul, Korea).
Change in whole body fat-free mass | Baseline (test and retest), week 7, week 13
  Fat-free body mass (kg) is measured at morning after overnight fasting by bioimpedance device (InBody 770, Biospace Co. Seoul, Korea)
Change in whole-body volume (cm^3) | Baseline (test and retest), week 7, week 13, before and after 6-weeks of ET.
  The 3D optical body (3DO) scan is used to measure whole-body volume, the volume of the body segments, and waist, hip, and thigh circumference. For 3DO, Fit3D ProScanner (Redwood City, CA, USA) is used.
Change in blood count determined from the venous blood sample obtained in the morning after overnight fasting before, mid, and after 12-week resistance training | Baseline (test and retest), week 7, week 13
  Full blood count is measured by hematology analyzer (Sysmex KX-21N, Sysmex Corp., Japan)
Change in C-reactive protein (CRP) determined from the venous blood sample obtained in the morning after overnight fasting before, mid, and after 12-week resistance training | Baseline, week 7, week 13
  Serum CRP is measured by high-sensitivity ELISA kit (Quantikine HS, R&D Systems, Minneapolis, USA).
Self-reported measure of physical activity | Baseline, week 13
  Investigated by the Global Physical Activity Questionnaire (GPAQ), a standardized 16-question questionnaire that assesses categories of low, moderate, and vigorous physical activity (in metabolic equivalent [MET] minutes per week) in three different domains: activity at work, travel to and from places, and leisure activities. Also, sedentary behavior (minutes per week) is assessed.
Sleep self-assessment | Baseline, week 13
  Investigated by The Pittsburgh Sleep Quality Index (PSQI) questionnaire which consists of questions of a four-point Likert scale (0-3), with higher scores representing greater sleep difficulties.
Self-report of eating disorder behaviors and attitudes | Baseline, week 13
  Investigated by the Eating Disorder Examination Questionnaire (EDE-Q), which assesses the extent, frequency, and severity of eating disorder-related behaviors on a seven-point Likert scale or occurrence over a 28-day period. Higher scores represent higher levels of eating disorders.
Self-estimated energy availability | Week 13
  Investigated by the Low Energy Availability Questionnaire (LEAF-Q for females, LEAM-Q for men) which identifies persons at risk for low energy availability by utilizing subsets of gastrointestinal symptoms, injury frequency, and menstrual dysfunction (in women). A score ≥8 indicates that an individual is at risk for low energy availability.
Self-measure of perceived stress | Baseline, week 7, week 13
  Investigated by Perceived Stress Scale (14 items); from 0 (never) to 4 (very often). The scores are obtained by reverse scoring the positively stated items (7 items) and then summing the points across all 14 items.
Recovery of muscle swelling after acute resistance exercise (RE) | Week 12: before and after the second last and the last training session, and once during the days in between
  The 3D optical body (3DO) scan is used to measure whole-body volume, the volume of the body segments, and waist, hip, and thigh circumference. For 3DO, Fit3D ProScanner (Redwood City, CA, USA) is used.
Recovery of muscle strength after acute resistance exercise (RE) | Week 12: before and after the second last and the last training session, and once during the days in between
  Maximal voluntary concentric muscle strength of leg extensors (kg) is determined in horizontal leg press device (David 210) via a one-repetition maximum (1RM) test. Maximum strength test is performed according to the NCSA guidelines.
Subjective muscle soreness after acute resistance exercise (RE) | Week 12: before the second last and the last training session, and once during the days in between
  Subjective muscle soreness is determined by a questionnaire and rated on a Likert scale of 0 (= no pain) to 5 (= maximum pain) for the overall muscle soreness of the quadriceps muscles during palpation of the muscle belly and walking up and down stairs, squatting, and sitting down.
Time to exhaustion (TTE) | Baseline, week 7 (post)
  TTE is the elapsed time from the beginning of the RAMP test to the point of test cessation. Test cessation is determined as the point at which the participant is unable to maintain a cadence above 60 rpm after one warning, despite heavy encouragement.
Change in maximal oxygen uptake | Baseline, week 7 (post)
  Maximal oxygen uptake (VO2max) is determined by expired gas analysis using breath-by-breath with a metabolic cart (Jaeger Vyntus TM CPX, CareFusion Germany 234 GmbH, Hoechberg, Germany) during an incremental RAMP test. VO2max is determined as the highest oxygen uptake over 30 seconds.
Change in the first ventilatory threshold | Baseline, week 7 (post)
  The first ventilatory threshold is determined by expired gas analysis using breath-by-breath with a metabolic cart (Jaeger Vyntus TM CPX, CareFusion Germany 234 GmbH, Hoechberg, Germany). The first ventilatory threshold is determined as the point during a RAMP test at which ventilatory equivalent (Ve/Vo2) begins to increase systematically. This point is determined graphically by plotting Ve/Vo2 onto the y-axis and oxygen consumption onto the x-axis.
Change in the second ventilatory threshold | Baseline, week 7 (post)
  The second ventilatory threshold is calculated by expired gas analysis using breath-by-breath with a metabolic cart (Jaeger Vyntus TM CPX, CareFusion Germany 234 GmbH, Hoechberg, Germany). The second ventilatory threshold is determined as the point during a RAMP test at which carbon dioxide equivalent (Ve/VCO2) begins to increase. This point is determined graphically by plotting Ve/VCO2 onto the y-axis, and oxygen consumption (ml/min/kg) to the x-axis.
Changes in cardiac output | Baseline, week 7 (post)
  Cardiac output will be measured with an impedance cardiograph (ICG) device (PhysioFlow, Manatec Biocmedical, Paris, France). ICG calculates cardiac output by calculating the change in transthoracic impedance during cardiac ejection, allowing the determination of stroke volume multiplied by heart rate also calculated by the ICG device.
Changes in stroke volume | Baseline, week 7 (post)
  Stroke volume will be measured with an impedance cardiograph (ICG) device (PhysioFlow, Manatec Biocmedical, Paris, France). Stroke volume is the amount of blood ejected from the ventricle with each cardiac cycle.
Changes in heart rate | Baseline, weeks 1-6 of ET, week 7 (post)
  Heart rate will be monitored continuously during both endurance testing, as well as endurance exercise sessions. The device used for heart rate monitoring is Polar Vantage V2 (Polar Electro Oy, Kempele, Finland) and heart rate will be assessed using a Polar H10 heart rate sensor (Polar Electro Oy, Kempele, Finland) attached with a chest wrap.
Changes in blood lactate concentration | Baseline, week 1 of ET, week 7 (post)
  Capillary blood samples will be taken from the fingertip after each movement economy interval, after an incremental RAMP test, and after the ET sessions during the first training week. Lactate concentrations (mmol/l) will be analysed with the EKF-diagnostics Biosen C-line device.
Changes in blood glucose concentration | Baseline, week 1 of ET, week 7 (post)
  Capillary blood samples will be taken from the fingertip after each movement economy interval, after an incremental RAMP test, and after ET sessions during the first training week. Glucose concentrations (mmol/l) will be analysed with the EKF-diagnostics Biosen C-line device.
Changes in hematocrit | Baseline, week 7 (post)
  Hematocrit, the relative amount of red blood cells in the blood (%), is measured from the blood samples taken from the fingertip using a hemoglobinometry (HemoCue Hb-801) device.
Changes in hemoglobin concentration | Baseline, week 7 (post)
  Hemoglobin concentrations (g/DL) are measured from the blood samples taken from the fingertip using a hemoglobinometry (HemoCue Hb-801) device.
Changes in respitatory exhange ratio (RER) | Baseline, week 7 (post)
  RER is calculated by dividing carbon dioxide (CO2) production by oxygen (O2) consumption, enabling the determination of relative utilization of aerobic adenosine triphosphate (ATP) production systems.
Changes in arterial oxygen saturation | Baseline, week 7 (post)
  Arterial oxygen saturation is calculated from an earlobe continuously during endurance testing, using a pulse oximeter.
Changes in subjective rating of perceived exertion (RPE) | Baseline, weeks 1-6 of ET, week 7 (post)
  RPE is determined with a modified scale of 0-10, in which 0 stands for no exertion and 10 for maximal exertion.
Aerobic threshold | Familiarization
  Aerobic threshold is determined as the 0.3 mmol/l increase in lactate concentrations from the lowest value, to estimate appropriate training loads for movement economy testing in baseline and post measurements.
Changes in movement economy | Baseline, week 7 (post)
  Movement economy is measured as the mean oxygen uptake relative to a given power (W) output. As the number of intervals is four in each movement economy test, loads will be increased after every interval. The load in the last interval is aimed to be below the aerobic threshold.
Blood pressure | Baseline, week 7 (post)
  Systolic and diastolic arterial pressure (mmHg) are measured with OMRON blood pressure monitor. Before measurement, participants are sitting still for 5 minutes. During measurement, participants are advised to sit still and avoid talking.
Changes in heart rate variability (HRV) | Baseline, week 7 (post)
  HRV, a variability in time intervals between R-R intervals, is determined with Polar Vantage V2 (Polar Electro Oy, Kempele, Finland) and Polar H10 heart rate sensors (Polar Electro Oy, Kempele, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Juha P Ahtiainen, Assoc.Prof., Principal Investigator — University of Jyväskylä, Faculty of Sport and Health Sciences
Locations (1):
- University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to juha.ahtiainen@jyu.fi